CLINICAL TRIAL: NCT01670864
Title: Promoting Smoking Cessation in the Community Via Quit to Win Contest 2012: Aa Cluster Randomized Controlled Trial of 18 Districts in Hong Kong
Brief Title: Promoting Smoking Cessation in the Community Via Quit to Win Contest 2012
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Sophia Siu-chee Chan, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QTW2012
Record Dates: First submitted 2012-08-17; First posted 2012-08-22 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Comparative Effectiveness Research; Community-Based Participatory Research

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Counseling group (Experimental): Study participants in the counseling group will receive a brief on-site face-to-face smoking cessation counseling from our trained smoking cessation counselor on the study site after signing the consent form. They will receive advice on quitting smoking and specific warning about the hazardous effects of smoking on health. A special designed health education card, based on the health education model, will be also provided to the participants. Additional telephone follow-up counseling (reminder) at 1-week & 1-month will be made to the participants in this group.
  Interventions: Behavioral: Counseling group
- SMS intervention group (Experimental): Study participants in the SMS group will receive SMS text messages on smoking cessation advice and warning on the hazardous effects of smoking on health. The participants will receive a total of 16 tailored SMS messages after recruitment.
  Interventions: Behavioral: SMS intervention group
- Control group (No Intervention): Study participants in the control group will not receive any quitting assistance other than the self-help materials from the recruitment sites.

INTERVENTIONS:
Behavioral: Counseling group — The content for the brief counseling group adopts a AWARD approach including asking the smoking habit, warning about the health risks associated with smoking, advising the smokers to quit, referring to specialized service, and repeating the above messages. A special designed health education card, based on the health education model, will be also provided to the participants. Additional telephone follow-up counseling (reminder) at 1-week & 1-month will be made to the participants in this group.
  Arms: Counseling group
Behavioral: SMS intervention group — The text messages are divided into two groups which target to smokers who are ready to quit and those who are not ready to quit. For smokers who are ready to quit, messages would be focused on practical advice and emotional support. For smokers who are not ready to quit, messages would be focused on motivating the smokers to have quit attempt.
  Arms: SMS intervention group

SUMMARY:
Background According to the report of Census & Statistics Department, there are still 659,300 daily smokers (11.1%) in Hong Kong and smoking kills over 7,000 people per year. The Quit and Win programme provided another opportunity to reach large group of smokers, and it aims to widespread quit attempts among smokers via incentives in order to boost up the number of quitters. Although such competitions appear to reach large cohorts of smokers, there is still insufficient evidence of its effectiveness in helping smokers to achieve complete cessation.

Aim This project aims to promote and evaluate community-based smoking cessation services through the Quit to Win Contest organised in the 18 districts of Hong Kong. The specific objectives of the study are (1) to build capacity in the community on smoking cessation through a training programme; (2) to empower the participated NGOs (a) to raise the awareness of smoking cessation in the community level; (b) to reach as many smokers as possible; (c) to arouse the interest of smokers to quit, through organizing the Quit to Win Contest; (3) to test the effectiveness of community-based on-site face-to-face counselling and Short Message Service (SMS) message vs. self-help booklet to assist current smokers to quit smoking; and (4) to build-up a community-based participatory research (CBPR) model in smoking cessation intervention at a district level in Hong Kong.

Methods A community-based participatory (CBP) approach, which is an effective way to engage public health researchers and community members (NGOs, other major stakeholders, and participants), will be used. Two domains of outcome will be assessed: (1) Effectiveness of smoking cessation interventions, (2) process evaluation of the recruitment activities including number of eligible participants and amount of publicity.

Procedure At the recruitment sites, after screening for eligibility of participants for the Quit to Win Contest, smoking counselor will measure eligible participant's level of carbon monoxide (CO) on expired air, and provide the self-help smoking cessation materials developed by the Hong Kong Council on Smoking and Health (COSH). Then the counselor will explain and invite the participants to join the cluster randomized controlled trial on smoking cessation intervention. Participants will be allocated to one of the groups of the smoking cessation intervention. 3- and 6-month follow-ups will be conducted

Hypothesis We hypothesize that the on-site brief smoking cessation advice will lead to significant increases in rates of smoking cessation in the intervention group than the control group (with the self-help materials only). Another hypothesis to be tested is that the intervention of sending SMS messages of smoking cessation advice is effective to increase the quit rate comparing to the control group.

DETAILED DESCRIPTION:
According to the report of Census & Statistics Department (2011a), there are still 659,300 daily smokers (11.1%) in Hong Kong and smoking kills over 7,000 people per year (Lam et al., 2001). Smoking also led to an annual medical cost, long-term care and productivity loss of US$688 million in 1998 (McGhee et al., 2006), which was equivalent to 0.6% of GDP in the region (Census & Statistics Department, 2011b). Smoking is addictive, and it is difficult for motivated smokers to quit without assistance. On the other hand, many smokers may not be ready to quit or wanted to quit on their own, and it is difficult to reach them.

The Quit and Win programme provided another opportunity to reach large group of smokers, and it aims to widespread quit attempts among smokers via incentives in order to boost up the number of quitters (Cahill & Perera, 2011). Although such competitions appear to reach large cohorts of smokers, there is still insufficient evidence of its effectiveness in helping smokers to achieve complete cessation (Cahill & Perera, 2009).

In 2009, we conducted a 3-armed randomized controlled trial to compare the effectiveness of two additional interventions of a 3-minute brief telephone advice (TEL group) and 8 of SMS messages (SMS group) to the usual care of smoking cessation self-help material (Control group) in the Quit to Win Contest 2009 [cite the final report]. More than one thousand participants were successfully recruited in a period of 2 months, with an overall self-reported quit rate of 21.6% among the contestants. However, no statistical significant evidence was found for the additional brief telephone advice or the SMS messages in increasing the quit rate. In 2010, we conducted another RCT on the Quit to Win Contest 2010 to compare the effectiveness of an on-site face-to-face brief smoking cessation advice vs. self-help materials (control) to achieve quit rate and changes in smoking behaviors. Once again, we recruited over one thousand participants during a period of 2.5 months. A higher quit rate was observed in the intervention group (18.4%) than the control group (13.8%) at 6-month follow-up, although it was marginally statistical insignificant (p = 0.08) (Wong et al., 2012). To conclude, both Quit to Win Contests in Hong Kong have successfully reached and captured the interest of a large number of smokers in the community who otherwise may not even think about quitting smoking. On the other hand, additional smoking cessation interventions seem to boost up the quit rate among smokers who joined the Quit to Win contest, and a dose-response relationship may appear among the additional interventions.

The theory of The Health Action Process Approach (HAPA) suggests that one's intention of behaviour change can be fostered by knowing that the new behaviour has positive outcomes as opposed to the negative outcomes that accompany the current behaviour; and planning (action planning and coping planning) serves as an operative mediator between intentions and behaviour (Schwarzer, 2008). Previous evidence has shown the applicability of the HAPA in changing people's health behaviours, e.g., physical exercise, breast self-examination, seat belt use, dietary behaviours, and dental flossing; and its generalizability has been confirmed by Schwarzer (2008). A theory-based health education card (pocket size), which was guided by the HAPA, will be developed and distributed to the participants as a reminder and like a 'homework assignment' to be completed at home, for the purpose of enhancing their intention and practice of the suggested behaviour (quitting smoking).

Short-Message Service (SMS) is one of the new methods of communication in the recent decade and an expanding number of studies were conducted in 2000s since it is in a self-help mode, inexpensive (in terms of manpower), can be readily disseminated, and available immediately upon request. Research evidences suggested that the SMS-delivered health intervention (including smoking cessation) have positive short-term outcomes (Fjeldsoe et al., 2009). Specifically, the intervention may increase the intention of quitting (Yu, 2010, Ybarra, 2011), but the use of such program was under-utilized (Andrews et al., 2012). In 2009, we conducted a RCT to test the additional effect of 8 SMS smoking cessation advice toward smokers who participated in a Quit to Win contest towards self-help material [cite the final report]. Although the results did not support the additional effect of SMS smoking cessation advice, it may due to the deficient number of SMS messages provided.

Community-Based Participatory Research (CBPR) is a partnership approach in a scientific research that involves the collaboration among community partners and academic researchers throughout the research process (Israel et al., 1998). It has been found effective in enhancing community input, building community capacity, and addressing barriers to health in study participants who have historically been underrepresented in research (Andrews et al., 2012, Horowitz et al., 2009). Community partners have the capability of managing a great deal of resources and manpower, and utilizing their network within the community, which are beneficial to a scientific research involving population-based interventions. To effectively raise the awareness of the contest and recruit as many participants as we can from the community, working with NGOs in the 18 Hong Kong districts with a CBPR model may be one possible way of program implementation.

The challenge of applying the CBPR model in the smoking cessation program is to equip the staffs from NGO about the related skills and knowledge, and maintain the quality of research process and intervention. Therefore, training programme and briefing session will be provided to the participated NGOs for the relevant knowledge transfer. In addition, process evaluation will be conducted throughout the recruitment and research process so that the quality and integrity of the effort by the involved NGOs can be monitored and evaluated.

Hence, we proposed to (1) test the effectiveness of an on-site face-to-face counseling using a theory-based health education model vs. SMS message vs. self-help materials to assist smokers who participate in the Quit to Win Contest 2012; (2) use a Community-Based Participatory Research (CBPR) model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 cigarette per day in the past 3 months
* Able to communicate in Cantonese and read Chinese
* Have a local network mobile phone
* Exhaled carbon monoxide (CO) 4 ppm or above, assessed by a validated CO smokerlyzer

Exclusion Criteria:

* Smokers who have difficulties (either physical or cognitive condition) to communicate
* Currently following other forms of smoking cessation programme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1193 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The self-reported 7-day point prevalence (pp) quit rate of smoking at 3 months | Three months
  Whether the participant has quitted smoking in the past seven days at the time point of 3 months

SECONDARY OUTCOMES:
Biochemical validated and self-reported smoking habit at 3 and 6 months | 3 and 6 months after recruitment
  * Test the cotinine level in the saliva provided by the participants
  * Self-reported quit rate at 6 months
  * Rate of smoking reduction by at least of half
  * Number of quit attempts at 3 and 6 months
Service output of the community-based smoking cessation intervention | Whole project
  Assessed by a Process Evaluation onsite observation form, and a series of checklists including participants record list, proposal and final report from NGOs. The components of process evaluation, including context, reach, dose delivered, dose received, fidelity and recruitment will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong SAR, China